CLINICAL TRIAL: NCT01724216
Title: Magnetic Resonance Imaging Using Innovative Pulse Sequences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 114-2012-GES-0014
Record Dates: First submitted 2012-11-07; First posted 2012-11-09 (Estimated); Results first posted 2014-09-02 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-10

CONDITIONS: Clinical Indication for a Head MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pulse sequence software (Experimental): The central aim of this study is to acquire a set of images and associated technical and clinical information to facilitate regulatory submission of the pulse sequences being studied by GEHC. Segment 1 allows to collect a minimum of 10 subjects then evaluate if additional scans/enrollment needed Segment 2 will allow an additional 90 subjects if data needed
  Interventions: Device: pulse sequences

INTERVENTIONS:
Device: pulse sequences — Collect in vivo human data to demonstrate neurological Magnetic Resonance Imaging of subjects using a pulse sequence
  Other Names: zero TE pulse sequences

SUMMARY:
The purpose of the study is to collect in vivo human image data to demonstrate neurological magnetic resonance imaging (MRI) of subjects using short pulse sequences.

DETAILED DESCRIPTION:
This is a single-site; open-label, prospective research Study involving human subjects. There will be no comparative efficacy or safety analysis and therefore no randomization

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age
* Subject must be willing and able to undergo verbal and written informed consent
* Subject must have a clinical indication for a head MRI with and without Gadolinium-based contrast agent administration

Exclusion Criteria:

* Subjects who have any of the conditions below at the time of the enrollment or scan session are excluded from this study. Further, should it be determined by study staff that an enrolled subject meets any of the conditions below during the course of the study, the subject will be removed from the study.

  * Any contraindication to an MRI scan per the policy of Spectrum Health
  * Any contraindication to administration of an MRI contrast agent per the policy of Spectrum Health
  * Off-label utilization of contrast agents administered for the subject's clinical exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark C DeLano, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with orders from their doctor for an MRI were screened from Spectrum Health's Neurology Department. The study coordinator contacts each subject that met the inclusion criteria. If the subject is interested to volunteer, a copy of the Informed Consent was sent and appointment scheduled. Seg. 1 enrolled 11 subjects; no Seg. 2 enrollment.
Pre-assignment Details: This is a single arm study.
Groups:
- Single Arm: Magnetic Resonance Images Collected Using Innovative Pulse Sequences :
Period: Overall Study
Arm/Group | Single Arm
Started | 11
Completed | 10
Not Completed | 1
Not completed — Scan was not completed | 1

BASELINE CHARACTERISTICS:
Population: images collected
Groups:
- Single Arm: Magnetic Resonance Image Collection Using Innovative Pulse Sequences
Arm/Group | Single Arm
Number analyzed (Participants) | 10
Age, Customized [Number; unit: participants with images collected]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex/Gender, Customized [Number; unit: participants with images collected] | NA — Gender was not a data point collected during the study.
Region of Enrollment [Number; unit: particpants with images collected]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Head Images Successfully Collected
Description: Collect head human images and associated technical and clinical information to demonstrate neurological magnetic resonance imaging of subjects using short pulse sequence.
Time Frame: 6-months
Measure: Number; unit: Images
Units Other Than Participants: Images
Groups:
- Single Arm: Magnetic Resonance Imaging Using Innovative Pulse Sequences :
Arm/Group | Single Arm
Number analyzed (Participants) | 10
Number analyzed (Images) | 10
Images | 10

ADVERSE EVENTS:
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No